CLINICAL TRIAL: NCT02026752
Title: Collection of Plasma Samples From Human Immunodeficiency Virus (HIV) Type 1 (HIV-1) Infected Individuals for the Clinical Evaluation of the Aptima HIV-1 Quant Dx Assay
Brief Title: Collection of Samples From HIV-1 Infected Individuals for Evaluation of the Aptima HIV-1 Assay
Status: Completed | Type: Observational
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: HIVQPS-US12-001; HIVQPS-US12-002 (Other: Gen-Probe); HIVQPS-US12-003 (Other: Gen-Probe); HIVQPS-US12-004 (Other: Gen-Probe)
Record Dates: First submitted 2013-12-31; First posted 2014-01-03 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Population

SUMMARY:
The objective is to obtain plasma samples from Human Immunodeficiency Virus Type 1 (HIV-1) infected individuals that have viral loads across the dynamic range of the Aptima HIV-1 assay. The plasma samples will be tested in a method comparison study to support the approval of the Aptima HIV-1 assay on Gen-Probe's Panther testing system. The objective of the method comparison study is to evaluate the clinical utility of the Aptima HIV-1 assay by comparing the results to the FDA-licensed COBAS assay (Roche Molecular Systems, Inc., Branchburg, New Jersey) in plasma samples that have viral loads across the dynamic range of the Aptima HIV-1 assay.

ELIGIBILITY:
Inclusion Criteria

* The subject has documented HIV infection
* The subject is at least 15 years of age at the time of enrollment
* For ART subjects, subject has documented HIV-1 RNA levels above the lower limit of quantitation of an FDA-approved assay in a sample collected in the past 90 days.
* The subject (and/or legally authorized representative, if allowed) is willing and able to provide written informed consent before providing a specimen (a minor will need the documented consent of his/her parent or legal guardian, unless the site has an institutional review board [IRB]-approved waiver for parental consent for minors).

Exclusion Criteria

* A potential subject will be ineligible for the study if the subject, clinician, or medical record reports any of the following:
* Subject's HIV disease stage and/or current ART status is unknown.
* It is unknown if current or previous ART was changed or stopped due to therapy failure.
* For non-ART subjects, subject was previously on ART in the past 30 days
* Subject already participated in this study and subject's previous sample(s) was provided and not withdrawn (ie, subject has an evaluable sample in the study)
* Subject has a history of illness that the principal investigator (PI) or designee considers could interfere with or affect the conduct, results, and/or completion of the study
* Subject has a history of illness that the PI or designee considers could create an unacceptable risk to the subject if enrolled in the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected male and female subjects ≥15 years of age who are attending participating US medical facilities will be eligible to enroll. Participating sites may include academic institutions with clinical divisions, infectious disease clinics, and other medical facilities such as sexually transmitted infection, HIV, and public health facilities
Sampling Method: Non-Probability Sample
Enrollment: 468 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Quantitative detection of HIV-1 RNA | single baseline visit
  Regression parameters (intercept and slope) will be estimated from method comparison analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Wait, Study Director — Director
Locations (9):
- United States (9):
  - Palmtree Clinical Research Inc, Palm Springs, California
  - UCSD - AnitViral Research Center (AVRC), San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Miami - AIDS Clinical Research Unit, Miami, Florida
  - Community AIDS Network, Sarasota, Florida
  - Wishard Health Services, Indianapolis, Indiana
  - Louisiana State University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Jacobi Medical Center, The Bronx, New York